CLINICAL TRIAL: NCT06771661
Title: Parents' Experience of Child Loss During Pregnancy or Birth - an Explorative, Sequential Mixed-methods Study
Brief Title: Parents' Experience of Child Loss During Pregnancy or Birth
Status: Recruiting | Type: Observational
Sponsor: Fritz Sterr (Other)
Responsible Party: Sponsor-Investigator, Fritz Sterr, Research associate, Deggendorf Institute of Technology, Faculty of Applied Healthcare Sciences
Organization: Deggendorf Institute of Technology, Faculty of Applied Healthcare Sciences (Other)
Other Study IDs: GEHBa-202409-V-237-R2
Record Dates: First submitted 2024-12-19; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Stillbirth and Fetal Death; Miscarriages; Experience
Keywords: Pregnancy loss; Child loss; Qualitative research; Mixed-methods; Experience; Need; Parents; Perinatal loss; Fetal death; Miscarriage; Stillbirth
MeSH Terms: conditions — Stillbirth; Fetal Death; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parents after intrauterine or perinatal child loss
  Interventions: Other: Workshops; Other: Focus group interviews; Other: Narrative interviews; Other: Delphi approach

INTERVENTIONS:
Other: Workshops — The investigators will conduct workshops with parents to get closer to the main topic.
Other: Focus group interviews — The investigators will conduct focus group interviews with parents on their needs before and during child loss.
Other: Narrative interviews — The investigators will conduct narrative interviews with parents to gain an in-depth understanding of their lived experience before and during the intrauterine or perinatal child loss.
Other: Delphi approach — The investigators will carry out a Delphi approach with parents to translate and confirm or revise the findings into treatment recommendations for healthcare professionals.

SUMMARY:
The investigators are conducting a participatory study with and for parents after child loss during pregnancy or birth. Their aim is to develop treatment recommendations for healthcare professional. These focus on question, how to deal with parents when experiencing child loss.

DETAILED DESCRIPTION:
The entire study is following a participatory approach and including parents after stillbirth in the research team. Along a co-creative design, the investigators planned a multistep-explorative mixed-methods study.

In detail, three key steps will be conducted. First, workshops and focus groups will be carried out to identify central needs of affected parents. Afterwards, one investigator will interview the parents narratively to gain an in-depth understanding of their experiencs. Finally, these findings will be summarized and translated into treatment recommendations for healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* German speaking
* Living in Austria, Germany or Switzerland
* Child loss during pregnancy or birth
* Child loss within last 12 months
* Legal capacity
* Voluntary participation

Exclusion Criteria:

* Loss of child after birth
* Not speaking and understanding German
* Not in a good mental condition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents (mothers, fathers) will be recruited that lost their child during pregnancy or birth in hospitals, at home or birth houses.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Parent's experience | During pregnancy and up to 7 days after birth
  The investigators are interested in parents' in-depth and lived experience before and during their intrauterine or perinatal child loss.

SECONDARY OUTCOMES:
Parents' subjective needs | During pregnancy and up to 7 days after birth
  In qualitative interviews, the subjective needs that parents developed before and during their intrauterine or perinatal child loss will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rester, Prof. Dr., Study Chair — Deggendorf Institute of Technology
Locations (1):
- Deggendorf Institute of Technology, Faculty of Applied Healthcare Sciences, Deggendorf, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
The data to be collected is particularly sensitive and is stored securely and deleted after the study. Individual pseudonymised excerpts are made public in the publications.

REFERENCES:
- See also: Landing Page of the Study — https://www.th-deg.de/sterneneltern